CLINICAL TRIAL: NCT04716192
Title: Effects of Positional Release Technique on Pain, Range of Motion and Function in Patients With Unilateral Subacute Trapezitis
Brief Title: Positional Release Technique in Patients With Unilateral Subacute Trapezitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/20/1039 Sana Naz
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Cervical Spine Disease
Keywords: Positional release therapy; trapezitis; subacute, pain; cervical ROM
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional release technique (Experimental): Positional release technique, Mayofascial release technique and ultrasound
  Interventions: Other: Positional release technique; Other: Myofascial release technique & Ultrasound
- Mayofascial release technique and ultrasound (Active Comparator): Mayofascial release technique and ultrasound
  Interventions: Other: Myofascial release technique & Ultrasound

INTERVENTIONS:
Other: Positional release technique — Positional Release Technique The subject lies supine with therapist standing on the affected side; tender points are located along the upper fibres of the trapezius. Pressure will applied by pinching the muscle between the thumb and fingers. The subject's head is laterally flexed toward the side of tender point, then therapist grasps the subject's forearm and abducts shoulder to approximately 90° a slight flexion or extension is added to obtain fine-tune. The ideal position of comfort achieved is held for a period of 90 seconds and followed by a passive return of the body part to an anatomically neutral position continued for 5 minutes.
  Mayofascial Release Technique Therapeutic Ultrasound
  Arms: Positional release technique
Other: Myofascial release technique & Ultrasound — Myofascial Release Technique
  * Position of the patient - sitting comfortably with supported back, elbow flexed with forearm placed on a pillow. A low load, long duration stretch is applied along the lines of maximal fascial restrictions. The fascia is palpated and the pressure is applied directly to the skin, into the direction of restriction just until resistance (tissue barrier) is felt. The pressure will be applied for 90 to120 seconds. This procedure will carried out without sliding over the skin or forcing the tissue until the fascia complex starts to yield and a sensation of softening is achieved.
  * Therapeutic ultrasound with the frequency of 3Mhz , with continuous mode and an intensity of 0.1-1.5 W/cm2 for a duration of 5 min will given with the patient position back rest.

SUMMARY:
To assess the effects of positional release technique to improve the cervical range of motion, relieve pain and function in the patient with unilateral subacute trapezitis.

DETAILED DESCRIPTION:
Trapezius pain is the most common muscular pain due to increased stress which results in trapezitis. The trapezius muscle is postural muscle diamond shape highly susceptible to overuse. It helps in extension, neck rotation, and side bending. Trapezitis is frequently caused by bad posture, watching TV or working on computer for a long and use of thick pillo. Passive ROM may be painful and restricted due to protective spasm in muscle. This study will be a Randomized controlled study and will be conducted in Met Life Rehablitation center Lahore. The study will be completed within the time duration of six months . Consecutive sampling technique will be used to collect the data. The sample size of 44 patients will be taken in this study to find the effect of positional release technique in subacute unilateral trapezitis. Patient will be divided into two groups. Mayoficial release therapy and ultrasound will be given to both groups as a baseline treatment. (Group A will be treated with positional release technique, mayofascial release technique and ultrasound while Group B will be treated with mayofascial release technique and ultrasound). All measurements will be taken at baseline and at the end of 2nd week.Each group will be given 3 sessions per week for 2 weeks. Neck disability index will be used to measure function, Numeric pain rating scale will be used to measure pain intensity and goniometer will be used to measure cervical lateral flexion and extension and rotation range of motion. Data will be analyzed on SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Pain with less than 3 months duration
* Subjects of sub- acute trapezitis with trigger points
* Taut band palpable in upper trapezius muscle
* Excruciating spot tenderness at one point along the length of the taut band of the upper trapezius muscle
* Restriction in cervical lateral flexion when measured
* Pain increased by elongating (stretching) the trapezius muscle.

Exclusion Criteria:

* Traumatic Neck Injury
* Fracture of cervical vertebras
* Cervical Spinal Cord Compromise
* Cervical Radiculopathy
* Spondylolisthesis of the cervical spine
* A history of heart disease or the presence of a pacemaker

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-07-25 (Actual)

PRIMARY OUTCOMES:
UNIVERSAL GONIOMETER | 2 weeks
  UG is a reliable device to evaluate cervical ROM. The UG is cheap, easy to use, popular instrument and requires minimum training. Intra-rater reliability is observed for both raters measuring ACROM using UG, with ICC (2,1) ranging from 0.83 to 0.98.
NUMERIC PAIN RATING SCALE | 2 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes.
NECK DISABILITY INDEX | 2 weeks
  Methods of assessment for such disability, especially those targeted at activities of daily living which are most affected by neck pain, questionnaire 10-item scaled entitled the Neck Disability Index (NDI). Face validity was ensured through peer-review and patient feedback sessions. Test-retest reliability was conducted (Pearson's r = 0.89, p ≤ . 05)

CONTACTS AND LOCATIONS:
Overall Officials: Saima Zahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Met Life Rehab center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parab AA, Pattanshetty R. Effect of myofascial release versus muscle energy technique on trapezius spasm in head and neck cancer patients: A randomized clinical trial. Indian Journal of Physical Therapy and Research. 2019;1(2):114.
- [Background] Chaudhary ES, Shah N, Vyas N, Khuman R, Chavda D, Nambi G. Comparative study of myofascial release and cold pack in upper trapezius spasm. International Journal of Health Sciences & Research. 2013;3(12):20-7.
- [Background] Mishra D, Prakash RH, Mehta J, Dhaduk A. Comparative Study of Active Release Technique and Myofascial Release Technique in Treatment of Patients with Upper Trapezius Spasm. Journal of Clinical & Diagnostic Research. 2018;12(11).
- [Background] Karthick K. A Study on the Effectiveness of Positional Release Therapy in the Management of Trapezitis. Research & Reviews: Journal of Computational Biology. 2018;6(2):19-25.